CLINICAL TRIAL: NCT05710393
Title: Hidradenitis Suppurativa - a Mendelian Trait? Genetic Pedigree and Linkage Analysis
Brief Title: Hidradenitis - an Analysis of Genetic Traits and Linkages in Families
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB18-1861
Record Dates: First submitted 2023-01-25; First posted 2023-02-02 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; HS; Acne inversa; Abscess; Boils
MeSH Terms: conditions — Hidradenitis Suppurativa; Abscess; Furunculosis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood (adults, approx. 8-9 mL), (pediatric, 2-4 mL); or Saliva (1.5 - 2.0 mL) specimen for DNA (Gene panel) analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected: (Affected) persons with a medical history of symptoms related to Hidradenitis Suppurativa.
- Unaffected-control: (Unaffected) family of participants, having no history of symptoms related to Hidradenitis Suppurativa.

SUMMARY:
The aim of this study is to find a genetic link or family trait connecting persons with Hidradenitis Suppurativa (HS) to each other. As a result, discover the cause and perhaps treatment for Hidradenitis Suppurativa (HS).

DETAILED DESCRIPTION:
Hidradenitis suppurativa (HS) is a chronic, debilitating skin disease characterized by multiple abscesses located predominantly in areas such as armpit, genital, pelvic, and perineum. It is considered an orphan disease of unknown origin and no existing treatment with a population prevalence estimated between 1-4%. It develops in otherwise healthy patients after puberty and affects patients life-long. HS often requires multiple surgical procedures to drain large abscesses, or hospitalization to treat infected wounds, can lead to feelings of personal embarrassment and social stigmatization.

Anecdotal evidence from affected families shows that HS often "runs in families" and may be inherited in a Mendelian fashion; however, no adequately powered study has been undertaken to investigate this hypothesis. This project aims to characterize the inheritance pattern of HS in families, and identify the genetic cause of this disease in those families with evidence for monogenic inheritance.

Data collection includes blood sample analysis (DNA), medical history, and information pertaining to any known family history of HS, from which a familial pedigree can be generated. This 'family-based' genetic study design will include both affected and unaffected family members, ideally spanning several generations. Therefore, study patients will be asked to refer their immediate and extended (affected and unaffected) family members to this research study.

ELIGIBILITY:
Inclusion Criteria:

* Participants (affected) with Hidradenitis Suppurativa and related symptoms
* Family (unaffected) of participants with Hidradenitis Suppurativa

Exclusion Criteria:

* Children under 7-years of age

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with a history of Hidradenitis Suppurativa, and their biological family members.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-09-17 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Hidradenitis Suppurativa Genetic linkage | 1-Day Study Participation
  Determine the genetic linkage of Hidradenitis Suppurativa (HS). Measurements are based on Gene panel assays of DNA specimen (blood or saliva) to find rare variant(s) linked to HS. Specimen samples include those provided by affected participants, and when possible they're biological family.
  A Gene panel diagnostic determines the number of variants (or mutation) in multiple genes, potentially identifying a genetic linkage of mendelian inheritance.

SECONDARY OUTCOMES:
Demographics of Participant Population | 1-Day Study Participation
  Compare demographic variables of the affected population to analyze HS symptom history.
  Statistical Analysis of data collected via participant interview:
  Gender (at birth) Race (ethnicity) Age (at symptom start) Health history (related to HS) Family history (related to HS)
Pattern of Affected Family | 1-Day Study Participation
  Measure inheritance proximity pattern of biologically related family, affected by HS symptoms.
  A 'Pedigree' will be generated using family history data collected during the study interview:
  Immediate family - parental, sibling, children
  Extended family (paternal vs maternal) - uncle, aunt, cousin
  Outcomes could span multiple generations.
Number of Variants Shared | 1-Day Study Participation
  Determine the number of shared rare variants (or mutations) in genes associated with HS, between affected participants and their family. Measured by Gene panel assay of DNA specimen (blood or saliva)
  A Gene panel diagnostic determines the number of variants (or mutation) in multiple genes, potentially identifying a genetic linkage of mendelian inheritance.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nagele, MD, MSc, Principal Investigator — University of Chicago Medicine
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No